CLINICAL TRIAL: NCT03249948
Title: DOuble SEquential External Defibrillation for Refractory Ventricular Fibrillation - DOSE VF Pilot Study
Brief Title: DOuble SEquential External Defibrillation for Refractory VF Pilot Study
Acronym: DOSE-VF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Peel Regional Paramedic Service (Unknown); Toronto Paramedic Services (Unknown); Halton Region Paramedic Services (Other); County of Simcoe Paramedic Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DOSE-VF-PILOT
Record Dates: First submitted 2017-08-01; First posted 2017-08-15 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized study, with cluster units defined by EMS agency. Each cluster will crossover at three times during the one year trial so that each agency will spend 4 months in each arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard defibrillation (No Intervention): All defibrillation attempts will occur using the standard defibrillation method, i.e. defibrillation pads will be placed in the anterior-anterior configuration. The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
- Vector change defibrillation (Other): The first three shocks will occur with defibrillation pads placed in the anterior-anterior position. All further shocks will occur with the pads placed in the anterior-posterior position. The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
  Interventions: Procedure: Vector change defibrillation
- Double-sequential defibrillation (Other): The first three shocks will occur with defibrillation pads placed in the anterior-anterior position. For all further shocks, a second set of defibrillation pads (via a second on scene EMS or fire defibrillator) will be applied in the anterior-posterior position, and defibrillation will be carried out by sequential defibrillation shocks provided by the two defibrillators (i.e. with a short delay between the two defibrillators). The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
  Interventions: Procedure: Double-sequential defibrillation

INTERVENTIONS:
Procedure: Vector change defibrillation — Defibrillation using pad placement in anterior-posterior position.
  Arms: Vector change defibrillation
Procedure: Double-sequential defibrillation — Defibrillation using two defibrillators, one with pad placement in anterior-posterior position, and the other with pad placement in anterior-anterior position, delivering two rapid sequential shocks.
  Other Names: Double sequential external defibrillation; DSED
  Arms: Double-sequential defibrillation

SUMMARY:
Despite significant advances in resuscitation efforts, there are some patients who remain in refractory ventricular fibrillation (VF) during out-of-hospital cardiac arrest. Double sequential external defibrillation (DSED) and vector change defibrillation have been proposed as a viable option for patients in refractory VF. This pilot cluster randomized trial will compare (1) continued resuscitation using standard defibrillation; (2) resuscitation involving DSED; or (3) resuscitation involving vector change defibrillation, in patients presenting with refractory VF during out-of-hospital cardiac arrest. The results of this pilot study will provide critical data for planning a larger, adequately powered multi-site randomized controlled trial to clinically evaluate DSED and vector change defibrillation compared to standard therapy for patients in refractory VF.

DETAILED DESCRIPTION:
Double sequential external defibrillation (DSED) and vector change defibrillation have been proposed as viable options for patients in refractory ventricular fibrillation (VF) during out-of-hospital cardiac arrest. However, currently there is insufficient evidence to support a widespread implementation of this therapy. As such, a well-designed randomized controlled trial (RCT) employing a standardized approach to alternative defibrillation strategies early in the treatment of refractory VF is required to determine whether these treatments may impact clinical outcomes. This pilot cluster randomized trial will be conducted in the regions of Peel, Halton, Simcoe, and the city of Toronto, Ontario, Canada over a one year period of time. All adult (≥ 18 years) patients presenting in refractory VF (defined as patients presenting in VF and remaining in VF after three consecutive standard defibrillation attempts each separated by 2 minutes of CPR) during out-of-hospital cardiac arrest of presumed cardiac etiology will be assigned to be treated by one of three strategies: (1) continued resuscitation using standard defibrillation; (2) resuscitation involving DSED (two defibrillators, one using anterior-posterior pad placement and the second using anterior- anterior pad placement delivering two rapid sequential shocks for all subsequent defibrillation attempts, ± antiarrythmic use and epinephrine as per current provincial standard); or (3) resuscitation involving vector change (change of defibrillation pads from anterior-anterior to an anterior-posterior pad position) defibrillation. The cluster units will be defined by emergency medical service (EMS) agency and each cluster will crossover at three times during the trial so that each agency will spend 4 months in each arm of the study. Outcomes of interest will include return of spontaneous circulation (ROSC), termination of VF after the first interventional shock, termination of VF inclusive of all interventional shocks, and number of defibrillation attempts to obtain ROSC. The primary objectives of the pilot study are to determine the feasibility and required sample size of a full-scale RCT in this population.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, non-traumatic cardiac arrest of presumed cardiac etiology, presenting rhythm to EMS of ventricular fibrillation; no ROSC or non VF rhythm after three consecutive EMS shocks.

Exclusion Criteria:

* Traumatic cardiac arrest, patients with pre-existing do not resuscitate orders, presumed pregnancy, patients in recurrent ventricular fibrillation (defined as those with a secondary presentation of VF (not the presenting rhythm) or those presenting in VF but did not receive three consecutive defibrillation attempts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) | 1 day
  Binary outcome of whether or not patient returned to spontaneous circulation
Feasibility of double sequential external defibrillation | Day 1
  80% or greater of patients receiving proper randomization and 80% or greater receiving an intervention shock prior to shock 6

SECONDARY OUTCOMES:
VF termination after first interventional shock | 1 day
  Cessation of the VF waveform on defibrillator monitor at first rhythm analysis post interventional or standard shock. The interpretation will occur after three standard shocks have failed to terminate VF.
VF termination inclusive of all interventional shocks | 1 day
  Cessation of the VF waveform on defibrillator monitor at any rhythm analysis post interventional or standard shock. The interpretation will occur after three standard shocks have failed to terminate VF.
Number of defibrillation attempts to obtain ROSC | 1 day
  Total number of shocks required to achieve the first ROSC during resuscitation, inclusive of the first three standard shocks.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Cheskes, MD, Principal Investigator — Sunnybrook Centre for Prehospital Medicine
Locations (4):
- Canada (4):
  - Peel Regional Paramedic Service, Brampton, Ontario
  - Halton Region Paramedic Services, Oakville, Ontario
  - County of Simcoe Paramedic Services, Simcoe, Ontario
  - Toronto Paramedic Services, Toronto, Ontario